CLINICAL TRIAL: NCT03826303
Title: The Impact of Vaping Ethanol in the Evaluation of Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: U.S. Department of Justice (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: HM20015064; 2018-75-CX-0036 (Other Grant/Funding Number: Department of Justice)
Record Dates: First submitted 2019-01-30; First posted 2019-02-01 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Electronic Cigarette Use
MeSH Terms: conditions — Vaping | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- E-cigarette with ethanol, 1 puff (Experimental)
  Interventions: Other: E-cigarette liquid with ethanol, 1 puff
- E-cigarette without ethanol, 1 puff (Placebo Comparator)
  Interventions: Other: E-cigarette liquid without ethanol, 1 puff
- E-cigarette with ethanol, 10 puffs (Experimental)
  Interventions: Other: E-cigarette liquid with ethanol, 10 puffs
- E-cigarette without ethanol, 10 puffs (Placebo Comparator)
  Interventions: Other: E-cigarette liquid without ethanol, 10 puffs

INTERVENTIONS:
Other: E-cigarette liquid with ethanol, 1 puff — E-cigarette liquid with ethanol, 1 puff
  Arms: E-cigarette with ethanol, 1 puff
Other: E-cigarette liquid without ethanol, 1 puff — E-cigarette liquid without ethanol, 1 puff
  Arms: E-cigarette without ethanol, 1 puff
Other: E-cigarette liquid with ethanol, 10 puffs — E-cigarette liquid with ethanol, 10 puffs
  Arms: E-cigarette with ethanol, 10 puffs
Other: E-cigarette liquid without ethanol, 10 puffs — E-cigarette liquid without ethanol, 10 puffs
  Arms: E-cigarette without ethanol, 10 puffs

SUMMARY:
The purpose of this research study is to find out about ethanol-containing e-cigarettes impact ethanol breath tests, field sobriety tests, or other tests of sobriety. Ethanol is a common part of e-cigarette liquids.

ELIGIBILITY:
Inclusion Criteria:

* Individuals must be e-cigarette users who are 21-65, willing to provide informed consent, attend the lab sessions as needed. Participants must agree to use designated products according to study protocol.

Exclusion Criteria:

* Women will be excluded if they are breast-feeding or test positive for pregnancy (by urinalysis) at screening.
* Some study details about the eligibility criteria are purposely omitted at this time to preserve scientific integrity. Full details will be posted at the conclusion of the study.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-04-02 (Actual); Primary Completion 2022-04-08 (Actual); Study Completion 2022-04-08 (Actual)

PRIMARY OUTCOMES:
Preliminary breath test for ethanol | Conducted before and after the e-cigarette is used by the participant, at multiple time points (change from baseline reading at 27, 35, 40, 45, and 56 minutes after e-cigarette use)
  Initial type of breath test used (gives percent blood alcohol concentration)
Evidentiary breath test for ethanol | Conducted before and after the e-cigarette is used by the participant, at multiple time points (change from baseline at 29, 37, 42, 47, and 58 minutes after e-cigarette use)
  Secondary type of breath test used (gives percent blood alcohol concentration)
Standard Field Sobriety Test | Conducted before and after the e-cigarette is used by the participant, at multiple time points (change from baseline at 30 and 49 minutes after e-cigarette use)
  Test used to determine sobriety

OTHER OUTCOMES:
Direct Effects of Vaping Questionnaire | Administered after e-cigarette use (at 39 minutes after e-cigarette use)
  Questionnaire that asks participants about their vaping experience (10 questions, each scored from 0 - 100)
Biphasic Alcohol Effects Scale | Conducted before and after the e-cigarette is used by the participant (change from baseline at 39 and 54 minutes after e-cigarette use)
  Questionnaire that asks participants about effects associated with alcohol use (14 questions, each scored from 0 - 10)
General Labeled Magnitude Scale | Administered after e-cigarette use (at 39 minutes after e-cigarette use)
  Questionnaire that asks participants about flavor sensation, harshness/irritancy, and "throat hit" of the e-cigarette (3 questions, each scored from 0 - 100)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Breland, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-09-10): https://cdn.clinicaltrials.gov/large-docs/03/NCT03826303/ICF_000.pdf